CLINICAL TRIAL: NCT04447222
Title: COVID-19: Well-Being and HRQOL in Cancer Patients Who Participated in Prior Behavioral Clinical Trials
Brief Title: Impact of the COVID-19 Pandemic and HRQOL in Cancer Patients and Survivors
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0425; NCI-2020-03900 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0425 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-06-11; First posted 2020-06-25 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: COVID-19 Infection; Malignant Solid Neoplasm
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey): Participants complete a survey online over 35-45 minutes about their experiences regarding the COVID-19 pandemic.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Complete survey

SUMMARY:
This study uses questionnaires to gain an understanding of how experiences during the COVID-19 pandemic, regardless of COVID-19 status, may have impacted health-related quality of life (HRQOL) and other areas such as COVID-19-specific psychological distress, disruptions to health care, finances and social interactions in cancer patients. The coronavirus disease 2019 (COVID-19) is an infectious disease that is caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The information learned from this study will guide the development of psychosocial programs to improve patient care and outcomes in cancer patients and survivors in the context of facing a global pandemic.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess experiences during the coronavirus disease-2019 (COVID-19) pandemic (e.g., exposure, risk factors, testing, isolation, seropositivity, hospitalization, loss of family or friends); COVID-19-specific psychological distress (e.g., fear, anxiety and depressive symptoms); health, financial and social disruptions; perceived benefits and social support; and HRQoL and other psychosocial and behavioral factors in cancer survivors who participated in one of three prior clinical trials.

II. Evaluate the extent to which COVID-19 experiences are associated with COVID-19 specific psychological distress, health, financial and social disruptions, perceived benefits and social support, and HRQoL.

III. Evaluate the extent to which resiliency factors such as social support and perceived benefits assessed concurrently and other psychosocial measures assessed in the prior trials moderate the effects of COVID-19 experiences on COVID-19-specific psychological distress and HRQoL.

IV. Examine group differences in the outcomes assessed in the protocol relative to prior group assignment in the behavioral clinical trials.

OUTLINE:

Participants complete a survey online over 35-45 minutes about their experiences regarding the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Prior patients who participated in one of the following protocols: 2012-0112, 2009-0976, or 2005-0035
* Has an active email address or can be contacted via MyChart or personal email

Exclusion Criteria:

* No evidence of consent from prior clinical trials

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cancer who have participated in prior behavioral clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 1242 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Coronavirus disease-2019 (COVID19)-specific psychological distress | At baseline
  Assessed using a COVID-19 questionnaire. Responses are provided on a Likert scale (from 1 to 4) where participants are asked to rank statements from "strongly disagree" to "strongly agree.''
The extent to which COVID-19 experiences are associated with COVID-19 specific psychological distress, health, financial and social disruptions, perceived benefits and social support, and health-related quality of life (HRQoL) | At baseline
  Will be tested using path analysis. Path analyses also provides an opportunity to test direct and indirect or mediation effects. Significance and goodness of fit of the model will be interpreted using several indices. A Comparative Fit Index (CFI) value of 0.90 or greater and a Root Mean Square Error of Approximation (RMSEA) of 0.08 or less will be used to establish model fit. The Lagrange multiplier and the Wald tests will be used to guide model modifications.
Resiliency factors | At baseline
  Assessed using a COVID-19 questionnaire. Responses are provided on a Likert scale (from 1 to 4) where participants are asked to rank statements from "strongly disagree" to "strongly agree." The measure provides a total score summary that indicates the degree to which the COVID-19 pandemic has negatively impacted the participant. Items that tap into resiliency are reverse scored. Will use multigroup analyses by levels of the moderator to identify differences in the magnitude of the associations based on the level of the moderator.
Group differences in the outcomes assessed in the protocol relative to prior group assignment in the behavioral clinical trials | At baseline
  Will be assessed using appropriate analysis of covariance (ANCOVA) techniques adjusting for important confounders differentiating those who did and did not complete the current survey.
Health-related quality of life (HRQOL) | At baseline
  Assessed using the Functional Assessment of Cancer Therapy-7 (FACTG7). The FACTG7 is a well-validated and commonly used measure of HRQoL in oncology. A total score provides an index of HRQoL, with higher scores reflecting better HRQOL
General quality of life (QOL) | At baseline
  Will be assessed using the Medical Outcomes Study 36-item short-form survey (SF-36). The FACTG7 is a well-validated and commonly used measure of HRQoL in oncology. A total score provides an index of HRQoL, with higher scores reflecting better HRQOL
Sleep disturbances | At baseline
  Will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is an 18-item self-rated questionnaire that assesses quality of sleep and sleep disturbances over a 1-month period. The PSQI has good internal and test-retest reliability.
Depression | At baseline
  Will be assessed using the Centers for Epidemiological Studies-Depression measures (CES-D). The CES-D is a well-validated 20-item self-report measure of depression that focuses on affective components of depression. Internal consistency is high and it also has demonstrated adequate convergent validity with other measures of depression. Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Changes in anxiety | At baseline
  Will be assessed using the Speilberger State/Trait Anxiety Inventory (STAI). The STATE scale (Form Y-1) is a 20-item scale that provides information about a person's current level of anxiety. The TRAIT scale (Form Y-2) is a 20-item scale that provides information about a person's general anxiety. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80)
Perceived availability of social support | At baseline
  Will be measured using the 24-item Social Provisions Scale that includes subscales for attachment, social integration, opportunity for nurturance, reassurance of worth, reliable alliance, and guidance.
Elements of mindfulness | At baseline
  Will be assessed using the Five Facets of Mindfulness Questionnaire. This assessment provides statements relating to the five components observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience and asks participants to mark the extent to which each statement is true in their life, using a five-point scale.
Non-judgmental physical and emotional sensations associated with eating | At baseline
  Will be assessed using the Mindful Eating Questionnaire validated by Framson et al. at each time point. Scoring of this evaluation provides an overall "summary" score, as well individual scores in the five categories of awareness, distraction, dis-inhibition, emotions, and external factors while eating.
The degree to which participants exercise compassion towards themselves under difficult circumstances and how this impacts their emotions | At baseline
  Will be assessed using the Self-Compassion Scale. This assessment is a 12-item questionnaire that provides questions about self-judgments, self-kindness, common humanity, isolation, mindfulness and over-identification using a five-point scale.
Physical activity | At baseline
  Will be assessed with the Godin Leisure-Time Exercise Questionnaire. This questionnaire has been used extensively in research with cancer survivors. It is easy to administer. the activity score of 24 units and more as active (substantial benefits); the activity score of 14-23 units as moderately active (some benefits); and the activity score of 13 units and less as inactive (less substantial or low benefits) at first.
Intrusive thoughts, or the tendency to ruminate on or avoid thoughts about stressors | At baseline
  Will be measured using the Impact of Event Scale (IES) that assesses the two most common categories of responses to stressful events: intrusion (intrusively experienced ideas, images, feelings, or bad dreams) and avoidance (consciously recognized avoidance of certain ideas, feelings, or situations).
Basic fruit/vegetable intake | At baseline
  Will monitor patients' diets using The National Institutes of Health - Fruit and Vegetable Screener.
Usual intake of percentage energy from fat | At baseline
  Will be assessed using The National Institutes of Health - Fat Screener.
Engagement in the core mind-body practices that the patients learned | At baseline
  As engagement in mind-body practices has been found to decrease stress, engagement in the core Mind-body practices that the patients learned in the past will be assessed with an instrument that lists the different techniques and mind body practices and ask study participants how often they have practiced each technique. The scale goes from "not at all to more than once a day". The instrument also asks participants about the benefits obtained from practicing each technique, the scale goes from "does not apply/I did not practice to yes, definitively beneficial."

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org